CLINICAL TRIAL: NCT00442637
Title: Maintenance Treatment With Capecitabine and Bevacizumab Versus Observation After Induction Treatment With Chemotherapy and Bevacizumab as First-line Treatment in Patients With Advanced Colorectal Carcinoma
Brief Title: Maintenance Treatment Versus Observation After Induction in Advanced Colorectal Carcinoma
Acronym: CAIRO3
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dutch Colorectal Cancer Group (Other)
Collaborators: Koningin Wilhelmina Fonds (Other); Sanofi (Industry); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAIRO3
Record Dates: First submitted 2007-02-28; First posted 2007-03-02 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Colorectal Cancer Metastatic
Keywords: CAIRO3; DCCG; colorectal cancer; induction; metronomic chemotherapy; observation; capecitabine; bevacizumab; oxaliplatin
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; Bevacizumab; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): observation
  Interventions: Other: observation
- 2 (Active Comparator): capecitabine plus bevacizumab
  Interventions: Drug: capecitabine + bevacizumab

INTERVENTIONS:
Drug: capecitabine + bevacizumab — Ca 1250 mg/m2 daily orally continuously, B 7.5 mg/kg i.v. q 3 w
  Arms: 2
Other: observation — observation after induction treatment
  Arms: 1

SUMMARY:
The optimal duration of systemic treatment in patients with advanced colorectal cancer is unknown.

In this study the effects of bevacizumab and low-dose continuous chemotherapy with capecitabine is investigated in patients who have responded to 6 courses of oxaliplatin, capecitabine and bevacizumab ("induction treatment", at standard doses). This treatment is continued until progression or severe toxicity. This regimen is compared to the effects a observation without treatment after the induction treatment.

In case of disease progression, induction treatment will be reintroduced.

DETAILED DESCRIPTION:
Standard 1st-line treatment for patients with advanced colorectal cancer currently consists of chemotherapy plus bevacizumab. With this approach the median overall survival is approximately 20 months, and progression-free survival in first-line approximately 9-11 months. The optimal duration of treatment is unknown. Current data suggest that the efficacy of bevacizumab is dependent on concomitant use of chemotherapy. However, oxaliplatin almost invariably gives rise to neuropathy after 6-8 cycles. Prolonged use of capecitabine is associated with e.g. hand-foot syndrome. Lastly, the prolonged use of these agents is associated with considerable costs.

Evidence, mainly preclinical, suggests that continuous dosing metronomic chemotherapy may be more efficacious than interval-chemotherapy given at MTD. In this study the concept of metronomic chemotherapy is explored by administering a continuous daily instead of the usual 2 weeks-on/1 week-off oral dosing regimen of low-dose capecitabine plus bevacizumab as maintenance therapy after induction combination chemotherapy given at MTD plus bevacizumab.

ELIGIBILITY:
Before the start of induction therapy:

Inclusion Criteria:

* Histological proof of colorectal cancer (in case of a single metastasis, histological or cytological proof of this lesion should be obtained);
* Distant metastases (patients with only local recurrence are not eligible);
* Unidimensionally measurable disease (> 1 cm on spiral CT scan or > 2 cm on chest X-ray; liver ultrasound is not allowed). Serum CEA may not be used as a parameter for disease evaluation;
* In case of previous radiotherapy, at least one measurable lesion should be located outside the irradiated field.
* Ongoing or planned first line treatment with 6 cycles of Xeloda, Eloxatin, and Avastin.

Exclusion criteria

* Prior adjuvant treatment for stage II/III colorectal cancer ending within 6 months before the start of induction treatment
* Any prior adjuvant treatment after resection of distant metastases
* Previous systemic treatment for advanced disease

At randomisation:

Inclusion criteria:

* WHO performance status 0-1 (Karnofsky PS > 70%);
* Disease evaluation with proven SD, PR or CR according to RECIST after 6 cycles of MTD chemotherapy performed in week 3-4 of the 6th cycle induction therapy, and randomisation performed in week 3-5 of the 6th cycle (see time table);
* Laboratory values obtained ≤ 2 weeks prior to randomisation: adequate bone marrow function (Hb > 6.0 mmol/L, absolute neutrophil count > 1.5 x 109/L, platelets > 100 x 109/L), renal function (serum creatinine ≤ 1.5x ULN and creatinine clearance, Cockroft formula, > 30 ml/min), liver function (serum bilirubin ≤ 2 x ULN, serum transaminases ≤ 3 x ULN without presence of liver metastases or ≤ 5x ULN with presence of liver metastases);
* Life expectancy > 12 weeks;
* Age >= 18 yrs;
* Negative pregnancy test in women with childbearing potential;
* Expected adequacy of follow-up;
* Institutional Review Board approval;
* Written informed consent Exclusion criteria
* History or clinical signs/symptoms of CNS metastases;
* History of a second malignancy ≤ 5 years with the exception of adequately treated carcinoma of cervix or basal/squamous cell carcinoma of skin;
* Previous intolerance of XelodaR, EloxatinR, and/or AvastinR for which any of these drugs have been permanently discontinued; patients with previous dose reductions or delays are eligible; patients with grade 2 neurotoxicity after the 6th cycle are eligible, and retreatment with EloxatinR after PFS1 should depend on the grade of neurotoxicity at that moment;
* Known dihydropyrimidine dehydrogenase (DPD) deficiency;
* (Planned) radical resection of all metastatic disease;
* Uncontrolled hypertension, i.e. consistently > 150/100 mmHg;
* Use of more than 3 antihypertensive drugs;
* Significant cardiovascular disease < 1 yr before randomisation (symptomatic congestive heart failure, myocardial ischemia or infarction, unstable angina pectoris, serious uncontrolled cardiac arrhythmia, arterial thrombosis, cerebrovascular event, pulmonary embolism);
* Any of these significant cardiovascular events during previous fluoropyrimidine therapy;
* Chronic active infection;
* Any other concurrent severe or uncontrolled disease preventing the safe administration of study drugs;
* Any impairment of gastrointestinal function or -disease that may significantly impair the absorption of oral drugs (i.e. uncontrolled nausea, vomiting, diarrhoea (defined as >CTC grade 2), malabsorption syndrome, bowel obstruction, or inability to swallow tablets);
* Concomitant treatments: concomitant (or within 4 weeks before randomisation) administration of any other experimental drug under investigation; concurrent treatment with any other anti-cancer therapy; full-dose anticoagulation (is allowed if started during induction therapy);
* Continuous use of immunosuppressive agents (except the use of corticosteroids as anti-emetic prophylaxis/treatment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 635 (Estimated)
Dates: Start 2007-01; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival after re-introduction of MTD chemotherapy and bevacizumab (PFS2) | study duration

SECONDARY OUTCOMES:
Progression-free survival between observation versus maintenance therapy (PFS1) | study duration
Response rate during re-introduction of MTD chemotherapy and bevacizumab | study duration
Toxicity | study duration
Quality of life | study duration
Overall survival | study duration
Translational research | study duration

CONTACTS AND LOCATIONS:
Overall Officials: C. JA Punt, MD PhD, Principal Investigator — Amsterdam Medical Centre, Amsterdam Netherlands
Locations (1):
- University Medical Center Nijmegen, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] Kurk S, Peeters P, Stellato R, Dorresteijn B, de Jong P, Jourdan M, Creemers GJ, Erdkamp F, de Jongh F, Kint P, Simkens L, Tanis B, Tjin-A-Ton M, Van Der Velden A, Punt C, Koopman M, May A. Skeletal muscle mass loss and dose-limiting toxicities in metastatic colorectal cancer patients. J Cachexia Sarcopenia Muscle. 2019 Aug;10(4):803-813. doi: 10.1002/jcsm.12436. Epub 2019 May 15. PMID 31094083
- [Derived] Goey KKH, Elias SG, van Tinteren H, Lacle MM, Willems SM, Offerhaus GJA, de Leng WWJ, Strengman E, Ten Tije AJ, Creemers GM, van der Velden A, de Jongh FE, Erdkamp FLG, Tanis BC, Punt CJA, Koopman M. Maintenance treatment with capecitabine and bevacizumab versus observation in metastatic colorectal cancer: updated results and molecular subgroup analyses of the phase 3 CAIRO3 study. Ann Oncol. 2017 Sep 1;28(9):2128-2134. doi: 10.1093/annonc/mdx322. PMID 28911067
- [Derived] Simkens LH, van Tinteren H, May A, ten Tije AJ, Creemers GJ, Loosveld OJ, de Jongh FE, Erdkamp FL, Erjavec Z, van der Torren AM, Tol J, Braun HJ, Nieboer P, van der Hoeven JJ, Haasjes JG, Jansen RL, Wals J, Cats A, Derleyn VA, Honkoop AH, Mol L, Punt CJ, Koopman M. Maintenance treatment with capecitabine and bevacizumab in metastatic colorectal cancer (CAIRO3): a phase 3 randomised controlled trial of the Dutch Colorectal Cancer Group. Lancet. 2015 May 9;385(9980):1843-52. doi: 10.1016/S0140-6736(14)62004-3. Epub 2015 Apr 7. PMID 25862517
- See also: Dutch Colorectal Cancer Group — http://www.dccg.nl